CLINICAL TRIAL: NCT05994755
Title: Association Between Cardiac ARRHYTHMIAs and Glycemic Variability in Patient With Type 2 Diabetes Monitored Through FREEstyle Libre and Bluetooth Technology. (ARRHYTHMIA FREE)
Brief Title: Association Between Cardiac ARRHYTHMIAs and Glycemic Variability in Patient With Type 2 Diabetes Monitored Through FREEstyle Libre and Bluetooth Technology.
Acronym: ARRHYTHMIAFREE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Antonio Rapacciuolo (Other)
Responsible Party: Sponsor-Investigator, Antonio Rapacciuolo, Principal Investigator, Federico II University
Organization: Federico II University (Other)
Other Study IDs: v1.0 22042023
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Diabetes; Arrhythmias; Atrial Fibrillation; Heart Failure
Keywords: diabetes type II; cardiac arrhythmias
MeSH Terms: conditions — Diabetes Mellitus; Arrhythmias, Cardiac; Atrial Fibrillation; Heart Failure; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to investigate the association between hypoglycemia, glycemic variability and cardiac arrhythmias in patients with diabetes Type II (T2D) already implanted with implantable cardiac defibrillator (ICD) and monitored remotely through Bluetooth technology and CGM (continuous glucose monitoring).

DETAILED DESCRIPTION:
Studies have shown that, when diabetes is present, there is a 35% to 60% greater risk of developing atrial fibrillation (AF). Diabetic patients with AF had a 61% increase in total mortality, a 77% increase in cardiovascular death and a 68% increase in heart failure. The greatest risk with the combination of AF and Type 2 Diabetes Mellitus (T2D) is a 79% increase in thromboembolic risk, particularly stroke.Hypoglycemia, frequently asymptomatic, may lead to cardiac arrythmias and induce an increased risk of cardiovascular morbidity and mortality in patients with T2D.

However, these conclusions need to be tempered by the limitations of all studies available to date, making it difficult to determine the onset and burden of AF, especially when it is not a monitored end-point.Since prospective randomized trials would be unethical, future research should focus on establishing whether such a link exists by employing an observational design and taking advantage of modern tools for long-term, real-life monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Patient already wearing CIEDs (Implantable Cardiac Electronic Device) with Bluetooth technology
2. Diabetes Type II, no insulin-treated
3. Over 18 years of age
4. Patient in Sinus Rhythm at the time of the enrollment
5. Ability to provide informed consent for registry participation and be willing and able to comply with the protocol described evaluations

Exclusion Criteria:

1. Subject who is, or is expected to be inaccessible for follow-up
2. pregnancy
3. Patients with persistent and longstanding persistent AF

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with Type II Diabetes already implanted with ICD and monitored remotely through Bluetooth technology and CGM (continuous glucose monitoring).
Sampling Method: Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2023-10-30 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
association between hypoglycemia, glycemic variability and cardiac arrhythmias | 6 months
  Incidence of cardiac arrhythmias (atrial fibrillation, atrial flutter, PVC...) detected through remote monitoring and correlation with hypoglycemic episodes.

SECONDARY OUTCOMES:
association between hypoglycemia, glycemic variability and heart failure | 6 months
  The relationship between cardiovascular disease (heart failure and ischemic heart disease) at baseline and clinically relevant cardiovascular disease in relation to TBR and TAR.

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided